CLINICAL TRIAL: NCT03787355
Title: Clinical Evaluation of Vertical Inter-implant Papilla Height in Platform Matched Implants in Comparison to Morse Connection Abutments: A Randomized Controlled Clinical Trial
Brief Title: Clinical Evaluation of Vertical Inter-implant Papilla Height in Platform Matched Implants in Comparison to Morse Connection Abutments
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Nada Zazou, Principle Investigator, assistant Lecturer, Modern Sciences and Arts University (MSA)., Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PERIO7:4:85
Record Dates: First submitted 2018-07-21; First posted 2018-12-26 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Interimplant Mucosa

STUDY DESIGN:
Intervention Model Description: Intervention versus Control.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cone Morse Connection Implants (Experimental): 2 neighboring Morse connection Implants
  Interventions: Combination Product: Morse connection Implants
- platform matched implants (Active Comparator): 2 neighboring platform matched implants.
  Interventions: Combination Product: Morse connection Implants

INTERVENTIONS:
Combination Product: Morse connection Implants — 2 neighboring morse connection Implants of Zinedent - Strauman

SUMMARY:
The complete fill of the inter-implant mucosa is much more challenging between two implants, than single implants, and is considered to be unpredictable (Tymstra et al., 2011). However, previous clinical studies have pointed to a relationship between the inter-implant mucosa fill and the horizontal distance between two adjacent implants. In particular, a greater inter-implant bone loss and the absence of the inter-implant mucosa were noted when neighboring implants were not separated by more than 3 mm (Tarnow, Magner and Fletcher, 1992).

The implant-abutment connection may have an impact on the amount such inter-implant bone loss, with morse-taper (MT) abutments emerging from the central region of the implant allow additional thickness in the horizontal soft-tissue component. This might help reducing marginal bone remodeling during biological width formation. Moreover, the literature indicates that the peri-implant bone strain vary significantly with the type of implant-abutment connection. The conical interface of MT connections helps dissipating the forces to the fixture.

The aim of the study is to clinically investigate the fate of soft tissue and papilla following crown placement on neighboring morse cone implants versus non-platform switched implants denoting the fate of soft tissue and papilla.

DETAILED DESCRIPTION:
* Study is to be conducted in the Oral Medicine and Periodontology department, Faculty of Oral and Dental Medicine - Cairo University, Egypt.
* Patients are to be selected from the outpatient clinic of the department of Oral Medicine and Periodontology-Cairo University.

Intervention:

Clinical examination:

1. Evaluation of the patient's general condition of the oral cavity, to make sure it complies with the criteria required to be enrolled in the study in terms of oral hygiene, pathological conditions, occlusion and inter-arch space.
2. Evaluation of the periapical condition and crestal bone level using a periapical radiograph.
3. Evaluation of the soft tissue biotype by trans-gingival piercing using a periodontal probe.
4. Width of keratinized gingiva (measured by a periodontal probe from the gingival margin to the mucogingival junction). It is measured at three areas (mesial, midbuccal and distal).

SURGICAL PROTOCOL (T0):

* Patients meeting the inclusion criteria, CBCT analysis and extensive diagnosis is done to plan for treatment.
* After randomization patients are assigned to one of the two groups
* After profound anesthesia administration, a full thickness crestal flap is reflected, sequential osteotomy of the implant sites to the desired depth is performed with great care of interimplant distance maintenance to a 3-4mm.
* Implant insertion and confirmatory x-rays are performed.
* Gingival formers will be placed.
* Flap closure is performed with interrupted 4-0 polyproplene sutures.

Postoperative Care:

Postoperative medication -Administration of:

1. Anti-inflammatory drugs (NSAIDS; Ibuprofen 600mg three times daily for 5 days) (Francesco Pieri et al, 2012).
2. Antiseptic mouth rinse (0.12% Chlorhexidine oral rinse) will be prescribed starting from the second day for 60 seconds two times a day for 14 days (Jun Yu et al, 2015).

   -Patient self-care instructions:
3. Application of an ice bag to the treated area for the first 24 hours (Francesco Pieri et al, 2012).
4. The patients were instructed to gently brush the operated area starting from the second day with a soft brush using roll technique.

Scheduled time of re-entry for patients:

3 months for prosthesis fabrication.

Clinical Examinations:

At the 3-month (T1), 6-month (T2) and 12-month (T3), the following clinical parameters will be recorded at the implant sites: Interimplant vertical papilla height, pink esthestic score (PES), probing depth (PD), peri-implant mucosal height (PMH), bleeding on probing at six sites of each implant (mesiobuccal, buccal, distobuccal, distolingual, lingual, and mesiolingual), and width of buccal keratinized mucosa (KM) at the midbuccal surface of each implant.

KM will be recorded as the linear distance from the mucosal margin to the mucogingival line.

Radiographic Examination Radiographic examination will be performed immediately after the surgical procedure (T0), and at T1 and T3. Standard periapical radiographs will be taken using a digital imaging software system.

ELIGIBILITY:
Inclusion Criteria:

* Systemically healthy patients.
* Good oral hygiene.
* Missing minimum of two neighboring maxillary teeth with sufficient bucco-palatal bone of ≥ 6mm.
* Interimplant distance planned to be 3-4 mm.
* Patient acceptance of more than one year of follow up.

Exclusion Criteria:

* Vertically deficient ridges. (≤10 mm)
* Smokers.
* Pregnant females.
* Thin biotype

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-02-17 (Actual); Primary Completion 2026-01-15 (Actual); Study Completion 2026-01-15 (Actual)

PRIMARY OUTCOMES:
Vertical papilla height | 6,12 months from T0 (Implant insertion)
  Change will be measured using periodontal probe in millimeters,

SECONDARY OUTCOMES:
Pink esthetic score (PES) | 12 months from T0 (Implant insertion)
  Numerical Rating Score (Fürhauser et al, 2005)
Crestal bone resorption | T0 at the time of implant insertion, T1 at 3 months after implant insertion and at T3 at 12 months after implant insertion.
  Using digital X-ray, bone resorption will be measured using a software in mm.
Probing depth (PD) | 3, 6,12 months from T0 (Implant insertion)
  six sites of each implant (mesiobuccal, buccal, distobuccal, distolingual, lingual, and mesiolingual)
Bleeding on probing (BOP) | at T2 (6 months after implant insertion) and T3 (12 months after Implant Insertion).
  Binary, Using periodontal probe.
Width of buccal keratinized mucosa (KM) | 3, 6,12 months from T0 (Implant insertion)
  Measured at the midbuccal surface of each implant using periodontal probe in mm.
Patient satisfaction (cleaning, food impaction) | At T2 (6 months after implant insertion) and T3 (12 months after Implant Insertion).
  Measured using Numerical Rating Scale (NRS) (Kiyak et al, 1984)

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided